CLINICAL TRIAL: NCT05256355
Title: Competency-based Assessment in Musculoskeletal Ultrasound- a Validity Study
Brief Title: Competency-based Assessment in Musculoskeletal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Maya Dreier Carstensen, MD, PhD fellow, Principal investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-002
Record Dates: First submitted 2022-02-11; First posted 2022-02-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Diseases
Keywords: Training; Ultrasound; Medical education
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSUS novices (Other): Measurement of competence
  Interventions: Other: musculoskeletal ultrasound
- MSUS intermediates (Other): Measurement of competence
  Interventions: Other: musculoskeletal ultrasound
- MSUS experts (Other): Measurement of competence
  Interventions: Other: musculoskeletal ultrasound

INTERVENTIONS:
Other: musculoskeletal ultrasound — The participants will perform four MSUS examinations which are all videorecorded. All videos will be rated by two blinded raters using the OSAUS assessment tool.

SUMMARY:
Early diagnosis and rapid treatment initiation are of most importance to prevent joint damage in patients with arthritis. Musculoskeletal ultrasound (MSUS) is becoming an integrated part of rheumatology routine care and is more sensitive than clinical examination for detecting synovitis even in the early stage of disease.

However, MSUS is highly operator dependent and competences are needed to ensure correct image interpretation. Traditionally competences are evaluated on how many examinations the trainees have performed, but the gold standard has now shifted towards competency-based education where objective assessment tools are the key element. A previous study has developed a scale for assessment of ultrasound competence, The Objective Structured Assessment of Ultrasound skills (OSAUS). Although expert consensus supports evidence of content validity of the assessment instrument, it is not known if the OSAUS scale can discriminate differences in performance scores between different levels of MSUS experience in rheumatology in a reliable way.

ELIGIBILITY:
Inclusion Criteria:

* Physicians working at the rheumatology departments in Denmark:

  1. Novices: No or little experience with MSUS (less than 100 examinations).
  2. Intermediates: Participated and completed at least one formal ultrasound course and more than 100 examinations (less than 1000 MSUS examinations).
  3. Physicians with a long experience in MSUS doing the procedure almost daily and providing teaching and/or research within this field (more than 1000 examinations).

Exclusion Criteria:

* No informed consent
* Novices/Intermediates: extensive experience in MSUS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Performance score | Up to 12 months
  Competence score assessed by blinded raters using a generic skills assessment scale (OSAUS).

CONTACTS AND LOCATIONS:
Overall Officials: Stine Maya Carstensen, MD, Principal Investigator — Copenhagen Center for Arthritis Research, Center for Rheumatology and Spine Diseases, Centre for Head and Orthopaedics, Copenhagen University Hospital - Rigshospitalet Glostrup, Copenhagen, Denmark
Locations (1):
- Stine Carstensen, Glostrup Municipality, Denmark

REFERENCES:
- [Result] Tolsgaard MG, Todsen T, Sorensen JL, Ringsted C, Lorentzen T, Ottesen B, Tabor A. International multispecialty consensus on how to evaluate ultrasound competence: a Delphi consensus survey. PLoS One. 2013;8(2):e57687. doi: 10.1371/journal.pone.0057687. Epub 2013 Feb 28. PMID 23469051
- [Result] Brown AK, O'Connor PJ, Wakefield RJ, Roberts TE, Karim Z, Emery P. Practice, training, and assessment among experts performing musculoskeletal ultrasonography: toward the development of an international consensus of educational standards for ultrasonography for rheumatologists. Arthritis Rheum. 2004 Dec 15;51(6):1018-22. doi: 10.1002/art.20844. PMID 15593176
- [Result] Carstensen SMD, Terslev L, Jensen MP, Ostergaard M. Future use of musculoskeletal ultrasonography and magnetic resonance imaging in rheumatoid arthritis. Curr Opin Rheumatol. 2020 May;32(3):264-272. doi: 10.1097/BOR.0000000000000709. PMID 32205568
- [Result] Nayahangan LJ, Dietrich CF, Nielsen MB. Simulation-based training in ultrasound - where are we now? Ultraschall Med. 2021 Jun;42(3):240-244. doi: 10.1055/a-1352-5944. Epub 2021 Jun 15. No abstract available. PMID 34130348
- [Derived] Carstensen SMD, Just SA, Pfeiffer-Jensen M, Ostergaard M, Konge L, Terslev L. Solid validity evidence for two tools assessing competences in musculoskeletal ultrasound: a validity study. Rheumatology (Oxford). 2024 Mar 1;63(3):765-771. doi: 10.1093/rheumatology/kead286. PMID 37307078